# Consent Form

The Acute Influence of Proprioceptive Neuromuscular Facilitation on Cervical Proprioception and Range of Motion.

Date: 25/02/2019

NCT Number: NCT04045106

Prepared by:

Mohammad AL-Jallad

ISTANBUL/TURKEY



# Consent to Participate in a Research

| | The Acute Influence of Proprioceptive Neuromuscular Facilitation on Cervical | | | |
|---|---|---|---|---|
| Title of Study: | Proprioception, Range of Motion and Strength. | | | |
| Investigator: | | | | |
| C | | Physiotherapy and | | |
| Name: | Dept: | Rehabilitation | Phone: | |
| | | | | - |

#### Introduction

- You are being asked to be in a research study of a treatment approach in physiotherapy practice. This approach is widely used in many areas however it is not widely used for neck region therefore this study will test this approach on three aspects joint position sense, range of motion and muscle strength.
- We ask that you read this form and ask any questions that you may have before agreeing to be in the study.

# **Purpose of Study**

- The purpose of the study is to investigate the effects of two approaches of the same treatment technique on neck Proprioception (joint position sense), range of motion and strength of muscles around the neck.
- Ultimately, this research will be used for Master degree thesis and may be used in external publications.

# **Description of the Study Procedures**

- If you agree to be in this study, you will be asked to do the following things:
  - 1. First an assessor will see you to assess 1. neck joint position sense 2. neck ROM using a specific instrument 3. neck muscles strength using a device.
  - 2. for intervention part a physiotherapist will ask you to sit on a chair or lay on a treatment table to apply the treatment approach which will only involve your neck and upper body.
  - 3. We will take the assessment 2 times first before intervention second immediately after intervention.
  - 4. Assessment might take from 10 to 20 minutes.
  - 5. Treatment might take from 10-20 minutes.

Note: Assessment and intervention will involve direct physical contact, if you are uncomfortable with this please inform the investigator before signing this document.

#### Risks/Discomforts of Being in this Study

- There are no reasonably foreseeable (or expected) risks. There may be unknown risks.
- Due to the nature of the approach that works on muscles a slight discomfort might occur.

### **Confidentiality**

- This study is anonymous. We will not be collecting or retaining any information about your identity.
- The records of this study will be kept strictly confidential. Research records will be kept in a locked file, and all electronic information will be coded and secured using a password protected file. We will not include any information in any report we may publish that would make it possible to identify you.

# Right to Refuse or Withdraw

• The decision to participate in this study is entirely up to you. You may refuse to take part in the study *at any time* without affecting your relationship with the investigators of this study or the institution. You have the right not to answer any single question, as well as to withdraw completely from the interview at any point during the process; additionally, you have the right to request that the interviewer not use any of your interview material.

# **Right to Ask Questions and Report Concerns**

You have the right to ask questions about this research study and to have those questions answered by the investigator before, during or after the research. If you have any further questions about the study, at any time feel free to contact me, [mohammad aljallad] at [mohamed.jallad.pt@gmail.com] or by telephone at [05050524725]. If you like, a summary of the results of the study will be sent to you. If you have any problems or concerns that occur as a result of your participation, you can report them to the investigator at the number above.

#### Consent

• Your signature below indicates that you have decided to volunteer as a research participant for this study, and that you have read and understood the information provided above. You will be given a signed and dated copy of this form to keep, along with any other printed materials deemed necessary by the study investigators.

| Participant Name: | | |
|--------------------------|--------------------|-------|
| Participant's Signature: | | Date: |
| Researcher Name: | Mohammad Al-Jallad | |
| Researcher's Signature: | | Date: |
| Assessor Name: | Çiçek Duman | |
| Assessor's Signature: | | Date: |